CLINICAL TRIAL: NCT01636102
Title: A Phase II Open Label, Uncontrolled, Multicenter Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Influenza Vaccine (Agrippal®), Formulation 2012/2013, When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Subunit Trivalent Nonadjuvated Influenza Study Vaccine in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71_32S; 2012-000063-24 (EudraCT Number)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Human Influenza
Keywords: Influenza; Adults; Elderly; Immunology; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: Trivalent influenza virus vaccine (TIV)

INTERVENTIONS:
Biological: Trivalent influenza virus vaccine (TIV) — A single 0.5 mL dose of the study vaccine supplied in prefilled syringes and administered intramuscularly in the deltoid muscle of (preferably) the non dominant arm

SUMMARY:
To evaluate the safety of a single intramuscular (IM) injection of trivalent nonadjuvated influenza study vaccine, formulation 2012/2013, in adult and elderly subjects and the antibody response to each influenza vaccine antigen, as measured by single radial hemolysis (SRH) and hemagglutination inhibition (HI) at approximately 21 days postimmunization in adult and elderly subjects in compliance with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers of 18 years of age or older;
2. Individuals able to comply with all the study requirements;
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, could have interfered with the subject's ability to participate in the study.
2. Individuals with any serious chronic or acute disease (in the judgment of the investigator), including but not limited to:

   * Medically significant cancer (except for benign or localized skin cancer, cancer in remission for ≥10 years or localized prostate cancer that has been clinically stable for more than 2 years without treatment);
   * Medically significant advanced congestive heart failure (ie. NYHA class III and IV);
   * Chronic obstructive pulmonary disease (COPD; i.e., GOLD Stage III and IV);
   * Autoimmune disease (including rheumatoid arthritis, except for Hashimoto's thyroiditis that has been clinically stable for ≥5 years);
   * Diabetes mellitus type I;
   * Poorly controlled diabetes mellitus type II;
   * Advanced arteriosclerotic disease;
   * History of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (e.g., Down's syndrome);
   * Acute or progressive hepatic disease;
   * Acute or progressive renal disease;
   * Severe neurological (es. Guillain-Barré syndrome) or psychiatric disorder;
   * Severe asthma.
3. Individuals with history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g. to eggs or eggs product as well as ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate).
4. Individuals with known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:

   * receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study;
   * receipt of immunostimulants;
   * receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study;
   * suspected or known HIV infection or HIV-related disease.
5. Individuals with known or suspected history of drug or alcohol abuse.
6. Individuals with a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion could have interfered with the safety of the subject.
7. Individuals who were not able to comprehend and to follow all required study procedures for the whole period of the study.
8. Individuals with history or any illness that, in the opinion of the investigator, posed additional risk to the subjects due to participation in the study.
9. Individuals who within the past 6 months have:

   * had any laboratory confirmed seasonal or pandemic influenza disease;
   * received any seasonal or pandemic influenza vaccine.
10. Individuals who received any other vaccine within 4 weeks prior to enrollment in this study or who were planning to receive any vaccine during the study.
11. Individuals with any acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days.
12. Individuals who experienced fever (i.e., axillary temperature ≥38°C) within the last 3 days of intended study vaccination.
13. Individuals participating in any clinical trial with another investigational product 4 weeks prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
14. Individuals who were part of study personnel or close family members conducting this study.
15. BMI >35 kg/m2.
16. Females who were pregnant (confirmed by positive urine pregnancy test) or nursing (breastfeeding). Females of childbearing potential who refused to use an acceptable method of birth control for the whole duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (1):
- University Hospital Ghent, Center for Vaccinology, Prof.Dr. G Leroux Roels, Ghent, Ghent, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 1 site in Belgium.
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- 18-60 Y: Subjects ≥18 years to ≤60 years of age who received one TIV vaccination
- ≥61 Y: Subjects ≥61 years of age who received one TIV vaccination
Period: Overall Study
Arm/Group | 18-60 Y | ≥61 Y
Started | 63 | 63
Completed | 63 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18-60 Y | ≥61 Y | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (12.8) | 69.2 (5.7) | 53.6 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 26 | 65
  Male | 24 | 37 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved Seroconversion or Significant Increase in SRH Area Against Each of Three Vaccine Strains After One Vaccination of TIV
Description: Immunogenicity was measured as the percentage of subjects who achieved seroconversion or significant increase in single radial hemolysis (SRH) area, against each of three vaccine strains, three weeks after vaccination (day 22), evaluated using SRH assay.
  Seroconversion or significant increase in SRH area was defined as the percentage of subjects with a negative prevaccination serum (SRH area ≤4 mm2) to a postvaccination SRH area ≥25 mm2; or a significant increase in antibody titer from a non-negative prevaccination serum, i.e., at least a 50% increase in area. The European (CHMP) criterion is met if percentage of subjects achieving seroconversion or significant increase in SRH area is >40% (≥18 years to ≤60 years) or 30% (≥61 years).
Time Frame: Day 22
Population: Analysis was done on the per-protocol (PP) set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | 18-60 Y | ≥61 Y
Number analyzed (Participants) | 62 | 62
Percentages of subjects
  A/H1N1 | 84 [72 to 92] | 53 [40 to 66]
  A/H3N2 | 81 [69 to 90] | 65 [51 to 76]
  B | 69 [56 to 80] | 73 [60 to 83]

2. Primary Outcome: Geometric Mean Ratio of Subjects Against Each of Three Vaccine Strains After One Vaccination of TIV
Description: Geometric mean ratio (GMR) of subjects was calculated as the ratio of postvaccination to prevaccination SRH geometric mean areas (GMAs), directed against each of three vaccine strains, three weeks after vaccination (day 22).
  The CHMP criterion was met if the geometric mean increase (GMR, day 22/day 1) in SRH antibody area is >2.5 (≥18 years to ≤60 years) or >2.0 (≥61 years).
Time Frame: Day 22
Population: Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | 18-60 Y | ≥61 Y
Number analyzed (Participants) | 62 | 62
Ratio
  A/H1N1 | 5.7 [4.3 to 7.55] | 2.88 [2.26 to 3.65]
  A/H3N2 | 5.52 [4.16 to 7.31] | 3.02 [2.35 to 3.86]
  B | 3.72 [2.69 to 5.15] | 4.06 [3.12 to 5.28]

3. Primary Outcome: Percentage of Subjects Who Achieved SRH Area ≥25 mm2 Against Each of Three Vaccine Strains After One Vaccination of TIV
Description: Immunogenicity was measured as the percentage of subjects achieving SRH area ≥25 mm2 against each of three vaccine strains at baseline (day 1) and three weeks after TIV vaccination (day 22).
  This criterion was met according to CHMP guideline if percentage of subjects achieving SRH area ≥25 mm2 is >70% (≥18 years to ≤60) or 60% (≥61 years).
Time Frame: Day 1 and 22
Population: Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- 18 - 60 Y: Subjects ≥18 years to ≤60 years of age who received one TIV vaccination
Arm/Group | 18 - 60 Y | ≥61 Y
Number analyzed (Participants) | 62 | 62
Percentages of subjects
  A/H1N1 (Day 1) | 34 [22 to 47] | 27 [17 to 40]
  A/H1N1 (Day 22) | 95 [87 to 99] | 71 [58 to 82]
  A/H3N2 (Day 1) | 23 [13 to 35] | 45 [32 to 58]
  A/H3N2 (Day 22) | 85 [74 to 93] | 92 [82 to 97]
  B (Day 1) | 61 [48 to 73] | 21 [12 to 33]
  B (Day 22) | 97 [89 to 100] | 82 [70 to 91]

4. Secondary Outcome: Numbers of Subjects Who Reported Solicited Local and Systemic Reactions (Day 1 - Day 4 Postvaccination)
Description: Safety was assessed as the number of subjects who reported solicited local and systemic reactions from day 1 up to and including day 4 after the TIV vaccination.
Time Frame: From day 1 through day 4 postvaccination
Population: Analysis was done on the safety dataset i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | 18-60 Y | ≥61 Y
Number analyzed (Participants) | 62 | 63
Number of subjects
  Injection site pain | 24 | 9
  Injection site ecchymosis | 0 | 1
  Injection site erythema | 3 | 4
  Injection site induration | 4 | 0
  Injection site swelling | 4 | 1
  Chills/shivering | 0 | 0
  Malaise | 2 | 1
  Myalgia | 5 | 3
  Arthralgia | 2 | 1
  Headache | 9 | 6
  Sweating | 3 | 2
  Fatigue | 8 | 3
  Body temperature (≥38°C) | 0 | 0

ADVERSE EVENTS:
Time Frame: From day 1 through day 22.
Description: Serious adverse events (SAEs) were collected from day 1 through day 22.
Arm/Group | 18-60 Y | ≥61 Y
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 28/63 | 18/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 18-60 Y (N=63) | ≥61 Y (N=63)
Fatigue (General disorders) | 8 | 3
Injection Site Erythema (General disorders) | 3 | 5
Injection Site Induration (General disorders) | 4 | 0
Injection Site Pain (General disorders) | 24 | 10
Injection Site Swelling (General disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Headache (Nervous system disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days